CLINICAL TRIAL: NCT06508411
Title: Exploration of the Relationship Between Sexual Health and Pain in the Context of Cancer in France: Cross-sectional Study
Brief Title: Exploration of the Relationship Between Sexual Health and Pain in the Context of Cancer in France
Acronym: CASEXPA
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2024 BALAYSSAC
Record Dates: First submitted 2024-07-08; First posted 2024-07-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2024-09

CONDITIONS: Pain; Cancer; Survivorship
Keywords: pain; neuropathic pain; sexual health; cancer patients; cancer survivors
MeSH Terms: conditions — Pain; Neoplasms; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- cancer patients and survivors: Individuals who self-identify as cancer patients or cancer survivors
  Interventions: Other: Pain screening

INTERVENTIONS:
Other: Pain screening — exploration of the relationship between pain and sexual health

SUMMARY:
The goal of this observational study is to explore the relationship between pain and sexual health in the context of cancer (cancer patients and cancer survivors). The main question it aims to answer is:

- Does pain interfere with sexual health in cancer patients and cancer survivors?

DETAILED DESCRIPTION:
Participants will be recruited through French cancer patient associations and will be invited to complete an online survey questionnaire, exploring:

* Sexual health and sexual satisfaction
* Pain severity and impact on daily activities
* Neuropathic pain
* Migraine
* Chemotherapy-induced peripheral neuropathy
* Quality of life, functioning, and symptoms
* Anxiety and depression
* Sociodemographic characteristics of patients
* Oncological characteristics

ELIGIBILITY:
Inclusion Criteria:

- Declaring themselves to be suffering from or having suffered from cancer recruited as such via appropriate communication systems (patient associations and social networks, etc.)

Exclusion Criteria:

* No command of the French language
* Residence outside France (verified with the department of residence in the questionnaire)
* Patient Companion
* Protected adult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male, female, non-binary
Study Population: Cancer patients and cancer survivors recruited via cancer patient associations
Sampling Method: Non-Probability Sample
Enrollment: 1661 (Actual)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
presence of pain | day 1
  BPI-SF questionnaire - Brief Pain Inventory short from (scores from 0 to 10 worse)
Sexual satisfaction | day 1
  SHQ-C22 questionnaire - Sexual Health Questionnaire (Scores from 0 to 100 better)

SECONDARY OUTCOMES:
Sexual satisfaction | day 1
  Visual analog scale (Scores from 0 to 10 better)
Quality of the sexual health | day 1
  SHQ-C22 questionnaire - Sexual Health Questionnaire (Scores from 0 to 100 better to worse depending of the items)
Pain severity and characteristics | day 1
  BPI-SF questionnaire - Brief Pain Inventory short from (scores from 0 to 10 worse)
Presence of neuropathic pain | day 1
  DN4 interview questionnaire - neuropathique pain 4 questions (scores from 0 to 7 worse)
Presence of migraine | day 1
  Items of the International Classification of Headache Disorders (typical headache that lasted 4-72 h without treatment, at least two of four typical headache characteristics (unilateral, pulsatile, pain intensity ≥4/10 on the visual analogue scale for pain, increase in pain with physical activity), at least one of two types of non pain-associated symptoms (nausea and/or vomiting, photophobia, and phonophobia))
Severity of chemotherapy-induced peripheral neuropathy (sensory and motor) | day 1
  QLQ-CIPN20 questionnaire - chemotherapy-induced peripheral neuropathy (scores from 0 to 100 worse)
Assessment of the quality of life | day 1
  QLQ-C30 questionnaire - quality of life questionnaire (scores from 0 to 100 better)
Assessment of the functioning dimensions | day 1
  QLQ-C30 questionnaire - quality of life questionnaire (scores from 0 to 100 better)
Assessment of the severity of symptoms | day 1
  QLQ-C30 questionnaire - quality of life questionnaire (scores from 0 to 100 worse)
Sociodemographic characteristics - age of patients | day 1
  age (years)
Sociodemographic characteristics - gender | day 1
  male, female, non binary
Sociodemographic characteristics - body mass index | day 1
  body mass index (kg/m²)
Sociodemographic characteristics - use of alcohol, tobacco, e-cigarette, cannabis; | day 1
  use of alcohol, tobacco, e-cigarette, cannabis (yes / no, yearly, monthly, weekly, daily)
Sociodemographic characteristics - marital status | day 1
  married; Single with occasional partner; Single without occasional partner
Sociodemographic characteristics - socioprofesional status | day 1
  Farmer ; Artisan ; Merchants/entrepreneurs ; White-collar professionals ; Intermediate professions ; Employees ; Workers ; Retirees ; Unemployed individuals
Sociodemographic characteristics - living area | day 1
  French department of living
Oncological characteristics - past and/or ongoing treatment | day 1
  currently being treated for cancer ; treated for cancer (today in remission and completed cancer treatments) ; treated for cancer (today cancer still present and treatments against cancer stopped)
Oncological characteristics - type of cancer | day 1
  Breast ; Prostate ; Pulmonary ; Blood ; Gynecological ; Kidney ; Colorectal ; Others
Oncological characteristics - date of cancer diagnosis | day 1
  date (mm/yyyy)

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France